CLINICAL TRIAL: NCT03742713
Title: A Phase Ila Exploratory 2-stage Design Study of CPC634 (CriPec® Docetaxel) Monotherapy in Subjects With Platinum Resistant Ovarian Cancer.
Brief Title: Efficacy Study of CPC634 (CriPec® Docetaxel) in Platinum Resistant Ovarian Cancer
Acronym: CINOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cristal Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-CL02
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Cancer; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPC634 (CriPec® docetaxel) (Experimental): CPC634 (CriPec® docetaxel) administered intra-venously every 21 days at 60 mg/m2
  Interventions: Drug: CPC634 (CriPec® docetaxel)

INTERVENTIONS:
Drug: CPC634 (CriPec® docetaxel) — Docetaxel containing CriPec® nanoparticles

SUMMARY:
The purpose of this study is to determine whether CPC634 (CriPec® docetaxel) is effective in the treatment of patients with advanced epithelial ovarian cancer who are resistant to prior platinum-based chemotherapy

.

DETAILED DESCRIPTION:
This Phase IIa exploratory 2-stage trial assessed the efficacy, safety and tolerability of CPC634 (CriPec® docetaxel) administered IV, Q3W to 25 subjects (13 in Stage 1 and 12 in Stage 2) with ovarian cancer that is resistant to prior platinum-based therapy. Subjects will be treated continuously every 21 days at 60 mg/m2, which is the RP2D of CPC634 (CriPec® docetaxel) that was determined in the Phase I CT-CL01, until disease progression, unacceptable toxicity, or discontinuation for any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 years.
2. Histologically or cytologically confirmed diagnosis of epithelial ovarian, fallopian or peritoneal cancer.
3. Platinum-resistant recurrent epithelial ovarian cancer (defined as progression within 6 months after last platinum dose). Subjects who have received a maximum of 2 prior treatment lines of which one could have been taxane- based.
4. Measurable disease according to RECIST version 1.1. Only CA-125 progression without any clinical or radiological progression is not allowed.
5. Performance status (WHO scale/ECOG) 1.
6. Estimated life expectancy of at least 5 months.
7. Toxicities incurred as a result of previous anti-cancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ Grade 2 (as defined by NCI- CTCAE version 5.0).
8. ANC ≥ 1.5 x 109/L; platelets ≥100 x 109/L; hemoglobin ≥ 5.58 mmol/L (≥ 9.00 g/dL)
9. Creatinine ≤ 1.75 x Upper Limit of Normal (ULN) and estimated creatinine clearance ≥ 30 mL/min according to Cockcroft-Gault formula; Serum albumin levels > 25g/L.
10. Serum bilirubin ≤ 1.5 x ULN except for subjects with Will Gilbert's syndrome; alkaline phosphatase, ASAT and ALAT ≤ 2.5 x ULN, unless related to liver metastases, in which case ≤ 5 x ULN is allowed.
11. Written informed consent according to local guidelines.

Exclusion Criteria:

1. Subjects with platinum-refractory disease. Refractory disease is defined by subjects who progressed during the preceding treatment or within 4 weeks after last dose of platinum containing therapy.
2. Less than four weeks since the last treatment with other anti-cancer therapies, (i.e. endocrine therapy, immunotherapy, radiotherapy, chemotherapy, etc.); less than eight weeks for cranial radiotherapy, and less than six weeks for nitrosoureas and mitomycin C prior to first study treatment.
3. Current or recent (within 28 days of first study treatment) treatment with another investigational drug or participation in another investigational study.
4. Active or symptomatic brain metastases. Subjects must be on a stable or decreasing dose of corticosteroids and/or have no requirement for anticonvulsants for five days prior to Cycle 1 day1 (C1D1).
5. Current malignancies other than epithelial ovarian, fallopian or peritoneal cancer, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
6. Major surgical procedure (including open biopsy, excluding central line IV and portacath) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.
7. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100mm Hg).
8. Grade ≥ 2 motor or sensory neuropathy symptoms (as defined by CTCAE version 5.0).
9. Known hypersensitivity to any of the study drugs or excipients or taxanes.
10. Any skin toxicity in the medical history of the subject of Grade ≥ 2 associated with impaired skin integrity (skin toxicity defined as any form of rash, HFS, skin ulceration, toxic epidermal necrolysis, eczema) or any skin toxicity for which systemic treatment was needed.
11. Clinically significant (i.e. active) cardiovascular disease defined as stroke, transient ischemic attack (TIA) or myocardial infarction within ≤ 6 months prior to first trial treatment.
12. Subjects, who are pregnant or breastfeeding. Serum pregnancy test to be performed within 7 days prior to study treatment start in subjects of childbearing potential.
13. Absence of highly effective method of contraception as of C1D1 in female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile).
14. Known hypersensitivity to dexamethasone or any other reason that would make the subject not eligible to receive dexamethasone.
15. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, drug or alcohol abuse, physical examination or laboratory findings) that may interfere with the planned treatment, affect subject compliance or place the subject at high risk from treatment- related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end of Cycle 6 (each cycle is 21 days)
  To determine the Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 of CPC634 (CriPec® docetaxel) monotherapy in subjects with ovarian cancer who are resistant to prior platinum-based therapy.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | At the end of Cycle 6 (each cycle is 21 days)
  To evaluate the incidence of Treatment-Emergent Adverse Events (safety and tolerability) of CPC634 (CriPec® docetaxel) according to NCI-CTCAE criteria (version 5.0)
Progression free survival | After 6 months
  Progression free survival (PFS) at 6 months based on RECIST version 1.1. and combined assessment using Gynecological Cancer Intergroup (GCIG) definitions for CA-125
GCIG CA-125 response criteria | At the end of Cycle 6 (each cycle is 21 days)
  GCIG CA-125 response criteria defined as at least a 50% reduction in CA-125 levels from a pretreatment sample confirmed and maintained for at least 28 days
Duration of response (DOR) | At the end of Cycle 6 (each cycle is 21 days)
  Duration of response (DOR) based on RECIST version 1.1 and combined assessment using GCIG definitions for CA-125
Time to progression (TTP) | After 6 months
  Time from treatment assignment to time of progressive disease per RECIST version 1.1.
Disease control rate (DCR) | At the end of Cycle 6 (each cycle is 21 days)
  Disease control rate (DCR) will be determined based on the percentage of subjects who have achieved complete response (CR), partial response (PR) and stable disease (SD) with treatment of CriPec® docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ledermann, MD,PhD, Principal Investigator — UCL Cancer Institute, London, UK
Locations (8):
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHU de Liège, Liège
- Netherlands (5):
  - University Medical Center Groningen, Groningen
  - Dijklander Hospital, Hoorn
  - Radboud University Medical Center, Nijmegen
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - Viecuri Medical Center, Venlo
- UCL Cancer Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No